CLINICAL TRIAL: NCT01695330
Title: A Phase II Study of Subcutaneous (SC) Bortezomib-Regimens for Patients With Relapsed/Refractory Multiple Myeloma (MM) Failing Prior Intravenous (IV) Bortezomib-Containing Regimens
Brief Title: Subcutaneous (SC) Bortezomib-Regimens for Patients With RR MM Failing Prior IV Bortezomib-Containing Regimens
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated by Sponsor of this study.
Sponsor: Oncotherapeutics (Industry)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X05384
Record Dates: First submitted 2012-08-24; First posted 2012-09-27 (Estimated); Results first posted 2017-01-16 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2016-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Relapsed; Refractory; Bortezomib; Subcutaneous; Oncotherapeutics
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Subcutaneous bortezomib (Experimental)
  Interventions: Drug: Subcutaneous bortezomib

INTERVENTIONS:
Drug: Subcutaneous bortezomib — Bortezomib will be administered SC at a dose of 1.0 mg/m2. Doses are to be administered on days 1, 4, 8, and 11 of a 28-day cycle. All other drugs used in combination with the SC bortezomib as well as their doses and schedules will be at the discretion of the Principal Investigator.
  Other Names: Velcade

SUMMARY:
This is a phase 2, multicenter, open label, nonrandomized study for patients with MM who will receive treatment with a SC bortezomib-containing combination regimen that does not contain thalidomide or vincristine. The patients will be required to have received a prior IV bortezomib containing combination regimen that did not contain thalidomide or vincristine and that differs from the SC bortezomib-containing one. In between the time that the patient received the IV bortezomib-based combination regimen and enrollment onto this study, patients may have received other non-bortezomib-based regimens as long as these treatments did not contain thalidomide or vincristine. This study will enroll patients who have relapsed or have become refractory to their prior IV-administered bortezomib-containing combination regimen as demonstrated by progressive disease while on or following that regimen. Patients must have received 4 doses of a minimum of 1.0 mg/m2 of bortezomib administered IV in no more than 4 weeks per cycle. Patients must have received at least one cycle meeting this definition and have shown progressive disease to be considered eligible. Patients who have relapsed or have become refractory to their most recent IV bortezomib-containing combination regimen are eligible regardless of when they received that regimen, as long as they meet the above criteria.

The study will consist of a screening period, followed by up to eight open label treatment cycles, a final assessment to occur 28 days after the end of the last treatment cycle, and a follow-up period.

DETAILED DESCRIPTION:
Primary Objectives:

• To establish the safety and tolerability of treatment with a SC bortezomib containing combination regimen for MM patients who have demonstrated progressive disease from a prior and different IV bortezomib containing combination regimen:

* To compare the incidence of PN between IV bortezomib and treatment with SC bortezomib in a subsequent anti-MM combination regimen
* To compare the severity of PN between IV bortezomib and treatment with SC bortezomib in a subsequent combination anti-MM regimen

Secondary Objectives:

* To compare the overall response rate [combined CR + very good partial response (VGPR) + PR + MR] following treatment with a SC bortezomib-containing combination regimen for MM patients who have demonstrated progressive disease from a prior and different IV bortezomib containing combination regimen
* To compare disease parameters following treatment with a SC bortezomib containing combination regimen for MM patients who have demonstrated progressive disease from a prior and different IV bortezomib containing combination regimen as follows:

  * time to progression
  * progression free survival
  * time to first response
  * duration of response
  * overall survival
* To determine the incidence and severity of injection-site reactions with SC administration of bortezomib

ELIGIBILITY:
Inclusion Criteria (Crit.):

1. Has a diagnosis of MM based on the following:

   Major crit.:
   1. plasmacytomas on tissue biopsy
   2. bone marrow plasmacytosis (> 30% plasma cells)
   3. m-spike on serum electrophoresis IgG > 3.5 g/dL or IgA > 2.0 g/dL; kappa or lambda light chain excretion > 1 g/day on 24 hour urine protein electrophoresis

   Minor crit.:
   1. bone marrow plasmacytosis (10% to 30% plasma cells)
   2. monoclonal Ig present but of lesser magnitude than given under major crit.
   3. lytic bone lesions
   4. normal IgM < 50 mg/dL, IgA < 100 mg/dL, or IgG < 600 mg/dL

   Any of the following sets of crit. will confirm the diagnosis of MM:
   * any 2 of the major crit.
   * major criterion 1 plus minor criterion 2, 3, or 4
   * major criterion 3 plus minor criterion 1 or 3
   * minor crit. 1, 2, and 3, or 1, 2, and 4
2. MM with measurable disease, defined as:

   * a m-spike on serum electrophoresis of at least 0.5 g/dL and/or
   * urine monoclonal protein levels of at least 200 mg/24 hours
   * for patients without measurable serum and urine M-protein levels, an abnormal free light chain ratio (normal value: 0.26 - 1.65)
3. Currently has progressive MM:

   * Relapsed following stabilization or a response to at least one IV bortezomib (bort.) containing combination regimen that did not contain thalidomide or vincristine or refractory defined as progressed while receiving that anti-myeloma tx
   * In between the IV bort.-based combination regimen and this study, the pt may have received other non-bort.-based regimens as long as these treatments did not contain thalidomide or vincristine
4. Voluntary written informed consent before performance of any study-related procedure not part of normal medical care
5. Age: ≥18 yrs at the time of consent
6. Able to adhere to the study visit schedule and other protocol requirements
7. ECOG performance status of ≤ 2 at study entry
8. Life-expectancy > 3 mos
9. Laboratory test results w/in these ranges at Screening and confirmed at enrollment prior to drug dosing on Cycle 1, Day 1:

   * ANC ≥ 1.5 x 109/L; if the bone marrow is extensively infiltrated (> 70% plasma cells) then ≥ 1.0 x 109/L
   * Platelet count ≥ 75 x 109/L; if the bone marrow is extensively infiltrated (> 70% plasma cells) then ≥ 50 x 109/L
   * Hgb > 8 g/dL
   * Calculated or measured CrCl of at least 30 mL/min. (see protocol)
   * Total Bili ≥ 1.5 x ULN
   * AST (SGOT) and ALT (SGPT) ≥ 3 x ULN ≥ 5 x ULN if hepatic metastases are present
   * Serum potassium WNL
10. Female pt is either postmenopausal for 1 year or greater before the screening visit, is surgically sterilized or if they are of childbearing potential, agree to practice 2 effective methods of contraception from the time of signing the informed consent form through 30 days after the last dose of VELCADE, or agree to completely abstain from heterosexual intercourse.
11. Male patients who agree to 1) practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug, or 2) completely abstain from heterosexual intercourse.

Exclusion Criteria:

1. POEMS syndrome
2. PCL
3. Primary amyloidosis
4. Diagnosed or treated for another malignancy w/in 3 yrs of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
5. ≤ Grade 2 peripheral neuropathy
6. Pt had myocardial infarction w/in 6 months prior to enrollment or has NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
7. Severe hypercalcemia, i.e., serum calcium ≤ 12 mg/dL (3.0 mmol/L) corrected for albumin
8. Undergone major surgery w/in 28 days prior enrollment or has not recovered from side effects of such therapy (see protocol)
9. Received the following prior therapy:

   * Thalidomide or vincristine alone or as part of a treatment regimen administered between the last IV bort.-based regimen and Cycle 1, Day 1 on this study. However, prior exposure to thalidomide or vincristine is allowed.
   * Chemotherapy w/in 21 days of study drugs (6 weeks for nitrosoureas)
   * Corticosteroids (>10 mg/day prednisone or equivalent) w/in 21 days of study drugs unless steroids are being administered at that dose or greater as part of the new regimen
   * Immunotherapy or antibody therapy as well as lenalidomide, arsenic trioxide or bort. w/in 21 days before study drugs
   * Radiation therapy w/in 21 days before study drugs. (see protocol for exceptions)
   * Use of any other experimental drug or therapy w/in 28 days of study drugs
10. Participation in clinical trials with other investigational agents not included in this trial, w/in 14 days of the start of this trial and throughout the duration of this trial.
11. Hypersensitivity to VELCADE (bort.), boron, or mannitol.
12. Concurrent use of other anti-cancer agents or treatments
13. Pregnant or lactating patients
14. Serious medical or psychiatric illness
15. Known positivity for HIV or hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R Berenson, MD, Principal Investigator — James R. Berenson, M.D., Inc.
Locations (1):
- James R. berenson, M.D., Inc., West Hollywood, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with MM who received treatment with a SC bortezomib-containing combination
Groups:
- Subcutaneous Bortezomib: patients with MM who received treatment with a SC bortezomib-containing combination. The patients were required to have received a prior IV bortezomib containing combination regimen that differs from the SC bortezomib-containing treatment.
- FG001: This is one-arm study.
Period: Overall Study
Arm/Group | Subcutaneous Bortezomib | FG001
Started | 52 | 0
Completed | 5 | 0
Not Completed | 47 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Subcutaneous Bortezomib
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Age, Continuous [Median (Standard Deviation); unit: years] | 62 (5.1)
Gender [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 5
The patients were required to have received a prior IV bortezomib containing combination regimen tha [Number; unit: participants] | 5

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective of This Study Will be to Investigate the Incidence and Severity of Peripheral Neuropathy Caused by a Prior Intravenous VELCADE-containing Regimen in Comparison to That Caused by a Subcutaneous VELCADE-containing Regimen.
Description: Definition of incidence: the number of participants enrolled in the study experiencing treatment-emergent peripheral neuropathy. Emergence of peripheral neuropathy is determined via neurological assessment conducted on Day 1 and Day 11 of each treatment cycle as well as during the End of Study visit.
  Definition of severity: the severity of any treatment-emergent peripheral neuropathy experienced by a patient on-study. Peripheral neuropathy severity is determined via neurological assessment conducted on Day 1 and Day 11 of each treatment cycle as well as the End of Study visit and is graded on a 0-4 scale based on CTCAE criteria.
  Incidence of Peripheral Neuropathy Definition: the number of participants enrolled in the study experiencing treatment-emergent peripheral neuropathy. Emergence of peripheral neuropathy is determined via neurological assessment conducted on Day 1 and Day 11 of each treatment cycle as well as during the End of Study visit.
Time Frame: Subjects eligible for this study will receive treatment with study drug for a maximum of eight 28 day treatment cycles.
Measure: Count of Participants; unit: Participants
Groups:
- Subcutaneous Bortezomib: Patients with MM who received treatment with a SC bortezomib-containing combination
Arm/Group | Subcutaneous Bortezomib
Number analyzed (Participants) | 5
Participants | 5

2. Secondary Outcome: Compare Overall Response Rate (CR + VGPR + PR + MR), Compare Disease Parameters, & Determine Incidence and Severity of Injection-site Reactions.
Description: Compare overall response rate [combined CR + very good partial response (VGPR) + PR + MR] and disease parameters [time to progression, -progression free survival, -time to first response, -duration of response, -overall survival] following treatment with a SC bortezomib-containing combination regimen for MM patients who have demonstrated progressive disease form a prior or different IV bortezomib-containing combination regimen. Determine incidence and severity of injection-site reactions with CS administration of bortezomib by number of patients with injection site reaction specific adverse events.
Time Frame: Subjects eligible for this study will receive treatment with study drug for a maximum of eight 28 day treatment cycles.
Reporting Status: Not Posted, anticipated posting 2017-10

ADVERSE EVENTS:
Groups:
- Subcutaneous Bortezomib: Bortezomib was administered SC at a dose of 1.0 mg/m2. Doses were administered on days 1, 4, 8, and 11 of a 28-day cycle. When administered subcutaneously, sites for each injection (thigh or abdomen) were rotated and reported. All other drugs used in combination with the SC bortezomib were recorded in the Case Report Forms along with their corresponding doses and schedules.
Arm/Group | Subcutaneous Bortezomib
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subcutaneous Bortezomib (N=5)
Gr3 Neturopenia (Immune system disorders) | 2 (2) — Neturopenia Gr3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No